CLINICAL TRIAL: NCT02618005
Title: Study for Evaluating the Impact of Continuous Consumption of Probiotics on Immune Function and Intestinal Microbiota in Astronauts Under Closed Microgravity Environment
Brief Title: Probiotics on Immune Function and Intestinal Microbiota in Astronauts Under Closed Microgravity Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yakult Honsha Co., LTD (Industry)
Collaborators: Japan Aerospace Exploration Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Probiotics
Record Dates: First submitted 2015-11-01; First posted 2015-12-01 (Estimated); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Immune Function and Intestinal Microbiota
Keywords: Astronauts; Probiotics; Immune function; Intestinal microbiota
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LcS group (Experimental): Consuming probiotic capsule
  Interventions: Dietary Supplement: Probiotic capsule
- Control group (No Intervention)

INTERVENTIONS:
Dietary Supplement: Probiotic capsule — Continuously take five capsules containing freeze-dried LcS on ISS for four weeks, from four weeks before the return (R-4W) to one day before the return (R-1d)
  Arms: LcS group

SUMMARY:
Human immune function and intestinal microbiota are suggested to be altered within long-duration stay in space. Accumulated evidences on earth support that Lacticaseibacillus paracasei strain Shirota (LcS) is a promising probiotic strain on improvement of immune function and intestinal microbiota. This study aims to investigate the impact of long-duration spaceflight as well as intake of LcS on the international space station (ISS), on immune system and intestinal microbiota in astronauts.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are scheduled to stay on the ISS for at least 3 months
* Individuals who fully understand the study protocol and provide written informed consent for the study participation

Exclusion Criteria:

* Individuals who routinely use antibiotic, laxative, and/or bowel regulating medicine
* Individuals who participate in other research that competes with this study in terms of the purpose and field, e.g., study with dietary management or intake of bifidobacteria/lactic acid bacteria, oligosaccharides, antibiotic, laxative, and/or bowel regulating medicine

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2022-04 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
Longitudinal changes in the number of LcS in feces | 9-18 months
  Number of LcS in feces will be assessed by PMA-qPCR, during pre-flight, in-flight and post-flight.
Longitudinal changes in the level of immune markers | 9-18 months
  Levels of immune markers in blood/saliva will be assessed by ELISA and bioassay, during pre-flight, in-flight and post-flight.
Longitudinal changes in numbers and composition of intestinal microbiota | 9-18 months
  Numbers and composition of bacteria in feces will be assessed by RT-qPCR/qPCR and next generation sequencer analysis, during pre-flight, in-flight and post-flight.

CONTACTS AND LOCATIONS:
Locations (1):
- Japan Aerospace Exploration Agency, Ibaraki, Japan